CLINICAL TRIAL: NCT03322046
Title: Heartmatters Challenge - First Responders
Acronym: HMC-FR
Status: Completed | Type: Observational
Sponsor: Boston Heart Diagnostics (Industry)
Collaborators: Heart Fit for Duty, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: CA-13-002
Record Dates: First submitted 2017-10-18; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Cardiovascular Diseases
Keywords: Therapeutic Lifestyle Change; Cardiovascular Disease; First Responders; Firefighters; CVD
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Therapeutic Lifestyle Change (TLC) Intervention Group: TLC group received CVD risk lecture, enrolled in lifestyle program, received follow-up visits from team practitioner after each blood draw, access to food journaling portal for 12 month period, telephonic coaching
  Interventions: Behavioral: Lifestyle Program
- Control Group: Control group received CVD risk lecture, then baseline, 3, 6, 12 month blood draws and 3 day food journals prior to each blood draw.

INTERVENTIONS:
Behavioral: Lifestyle Program — 4 elements: 1) Laboratory test results with diagnostic report describing results, 2) Lifestyle plan generated in online portal with personalized nutritional information based on combination of laboratory results and personal preferences, 3) online or smartphone food journaling application, 4) telephone based lifestyle coaching with Registered Dietitian.
  Groups: Therapeutic Lifestyle Change (TLC) Intervention Group

SUMMARY:
The purpose of this protocol is to observe whether providing the first responder population with a multi-tiered therapeutic lifestyle modification program, including regular blood testing, diet and telephonic lifestyle coaching, daily food journaling using web-based tools and smartphone apps can lead to positive changes in behavior, resulting in improvements in blood based markers of risk of cardiovascular disease (CVD) as well as improvements in weight and waist circumference.

DETAILED DESCRIPTION:
A cluster randomization of first responder communities in the metro Boston and metro Phoenix areas was performed. First responders attended a one hour lecture on the specific risks of CVD in that population and then qualified intervention candidates were enrolled into a lifestyle program, consisting of telephone-based coaching sessions with a registered dietitian and an online/app based food journaling program. Both groups had blood test draws at baseline, 3, 6 and 12 months. The intervention group met with the team practitioner to review results and progress after each blood draw. The test panel comprised blood-based markers of CVD risk associated with lipid metabolism, metabolics, inflammation and basic liver and kidney function.

ELIGIBILITY:
Inclusion Criteria:

1. Low apolipoprotein A-1 (apoA-1) levels in the very large alpha-1 HDL particle (<20 mg/dL for men, <30 mg/dL for women) OR increased waist size (at least 40 inches for men or 35 inches for women).
2. Internet access
3. 14 day food log completed prior to initiating the study intervention (or 3-day food log for the control group).

   -

Exclusion Criteria:

1. No insulin-requiring diabetes
2. No pregnancy or plans to get pregnant in next 12 months
3. Unable or unwilling to follow protocol
4. Unavailable for duration of study
5. Planning to change jobs during study term

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First responders: fire fighters, police officers, EMT personnel
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2013-10-08 (Actual); Primary Completion 2014-11-20 (Actual); Study Completion 2015-01-08 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 months
  Change in weight from baseline measurement
Reduction in waist circumference | 12 months
  Change in waist circumference from baseline measurement
Increase in large HDL subparticles | 12 months
  Change in concentration of large HDL particles measured by 2Dimensional gel electrophoresis

SECONDARY OUTCOMES:
Improvements in blood based markers of CVD risk | 12 months
  Markers involved in lipid metabolism, inflammation and metabolics

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dansinger, MD, Principal Investigator — Boston Heart Diagnostics
Locations (1):
- Boston Heart Diagnostics, Framingham, Massachusetts, United States

REFERENCES:
- [Result] Asztalos BF, Batista M, Horvath KV, Cox CE, Dallal GE, Morse JS, Brown GB, Schaefer EJ. Change in alpha1 HDL concentration predicts progression in coronary artery stenosis. Arterioscler Thromb Vasc Biol. 2003 May 1;23(5):847-52. doi: 10.1161/01.ATV.0000066133.32063.BB. Epub 2003 Mar 13. PMID 12637338
- [Result] Asztalos BF, Cupples LA, Demissie S, Horvath KV, Cox CE, Batista MC, Schaefer EJ. High-density lipoprotein subpopulation profile and coronary heart disease prevalence in male participants of the Framingham Offspring Study. Arterioscler Thromb Vasc Biol. 2004 Nov;24(11):2181-7. doi: 10.1161/01.ATV.0000146325.93749.a8. Epub 2004 Sep 23. PMID 15388521
- [Result] Kales SN, Soteriades ES, Christophi CA, Christiani DC. Emergency duties and deaths from heart disease among firefighters in the United States. N Engl J Med. 2007 Mar 22;356(12):1207-15. doi: 10.1056/NEJMoa060357. PMID 17377158
- [Result] Kales SN, Tsismenakis AJ, Zhang C, Soteriades ES. Blood pressure in firefighters, police officers, and other emergency responders. Am J Hypertens. 2009 Jan;22(1):11-20. doi: 10.1038/ajh.2008.296. Epub 2008 Oct 16. PMID 18927545
- [Result] Poston WS, Jitnarin N, Haddock CK, Jahnke SA, Tuley BC. The impact of surveillance on weight change and predictors of change in a population-based firefighter cohort. J Occup Environ Med. 2012 Aug;54(8):961-8. doi: 10.1097/JOM.0b013e31825296e0. PMID 22772954
- [Result] Schaefer EJ, Santos RD, Asztalos BF. Marked HDL deficiency and premature coronary heart disease. Curr Opin Lipidol. 2010 Aug;21(4):289-97. doi: 10.1097/MOL.0b013e32833c1ef6. PMID 20616715
- [Result] Soteriades ES, Hauser R, Kawachi I, Liarokapis D, Christiani DC, Kales SN. Obesity and cardiovascular disease risk factors in firefighters: a prospective cohort study. Obes Res. 2005 Oct;13(10):1756-63. doi: 10.1038/oby.2005.214. PMID 16286523
- [Derived] Gill R, Superko HR, McCarthy MM, Jack K, Jones B, Ghosh D, Richards S, Gleason JA, Williams PT, Dansinger M. Cardiovascular Risk Factor Reduction in First Responders Resulting From an Individualized Lifestyle and Blood Test Program: A Randomized Controlled Trial. J Occup Environ Med. 2019 Mar;61(3):183-189. doi: 10.1097/JOM.0000000000001490. PMID 30475306